CLINICAL TRIAL: NCT01468389
Title: A Randomized Multicenter Phase III Study:Taxanes or Platinum in Combination With Capecitabine Followed by Capecitabine Alone vs.Taxanes or Platinum Combined With Capecitabine in Advanced Adenocarcinoma of the Stomach or Esophagogastric Junction.
Brief Title: Taxanes or Platinum in Combination With Capecitabine Followed by Capecitabine Alone as First Line Treatment for Patients With Advanced Adenocarcinoma of Stomach or Esophagogastric Junction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Responsible Party: Principal Investigator, Xu jianming, The Affiliated Hospital of the Chinese Academy of Military Medical Sciences, The Affiliated Hospital of the Chinese Academy of Military Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGC001-307PLAH-XJM
Record Dates: First submitted 2011-11-04; First posted 2011-11-09 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; capecitabine; maintenance treatment
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Taxanes or Platinum in combination with Capecitabine (Active Comparator): The patients will received chemotherapy combining capecitabine with platinum or taxanes until progression.
  Interventions: Drug: Capecitabine
- chemotherapy followed by capecitabine alone (Experimental): The patients who has received 4 cycle chemotherapy combining capecitabine with platinum or taxanes and the result was SD or CR or PR,will be given capecitabine alone until progression.
  Interventions: Drug: capecitabine

INTERVENTIONS:
Drug: Capecitabine — 900-1000mg/m2 bid, days 1-14, every 3 weeks
  Arms: Taxanes or Platinum in combination with Capecitabine
Drug: capecitabine — Dosing schedule: 900-1000mg/m2 bid, days 1-14, every 3 weeks Maintenance dosing schedule: 1000-1250mg/m2 bid, days 1-14, every 3 weeks
  Arms: chemotherapy followed by capecitabine alone

SUMMARY:
The purpose of this study is to investigate whether Taxanes or Platinum Plus Capecitabine With Capecitabine Maintenance Treatment as 1st line treatment in he advanced gastric cancer is effective and safe.

ELIGIBILITY:
Inclusion Criteria:

1. Having signed informed consent
2. Age≥ 18 years old
3. Histologically confirmed gastric adenocarcinoma
4. Unresectable recurrent or metastatic disease
5. Previous neo-adjuvant or adjuvant treatment for gastric cancer, if applicable, more than 6 months
6. Previous chemotherapy with oxaliplatin or cisplatin or paclitaxel or docetaxel, if applicable, more than 12 months.
7. Measurable disease according to the RECIST criteria
8. ECOG performance status ≤2
9. Life expectancy of ≥3 month
10. No prior radiotherapy except radiotherapy at non-target lesion of the study more than 4 weeks
11. ALT and AST≤2.5 times ULN (≤5 times ULN in patients with liver metastases) Serum albumin level ≥3.0g/dL Serum creatinine ≤1.5ULN Bilirubin level ≤ 1.5 ULN WBC>3,000/mm3, absolute neutrophil count ≥1500/mm3, platelet>90,000/mm3, Hb>8g/dl

Exclusion Criteria:

1. Brain metastasis (known or suspected)
2. Previous systemic therapy for metastatic gastric cancer
3. Inability to take oral medication
4. Previous therapy targeting at angiogenesis or vasculogenesis pathway or other targeted therapy
5. Surgery (excluding diagnostic biopsy) within 4 weeks prior to study entry
6. Allergic constitution or allergic history to any investigating agents.
7. Severe heart disease or such history as recorded congestive heart failure, uncontrolled cardiac arrhythmia, angina pectoris needing medication, cardiac valve disease, severe abnormal ECG findings, cardiac infarction , or retractable hypertension.
8. Pregnancy or lactation period
9. Any investigational agent within the past 28 days
10. Other previous malignancy within 5 year
11. Pre-existing neuropathy>grade 1
12. Legal incapacity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-01 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 1 year

SECONDARY OUTCOMES:
Tumor response rate | 1 year
disease control rate | 1 year
overall survival | 3 year
adverse events | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Xu jianming, M.D., Principal Investigator — The Affiliated Hospital of the Chinese Academy of Military Medical Science
Locations (1):
- 307 Hospital of PLA, Beijing, Beijing Municipality, China